CLINICAL TRIAL: NCT04823390
Title: Anesthetist Controlled Versus Patient-controlled Sedation: Risks and Benefits, a Randomized Controlled Trial
Brief Title: Anesthetist Controlled Versus Patient-controlled Sedation: Risks and Benefits
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Shamma, Assistant lecturer of anaesthesia, surgical ICU and pain management kasr al aini, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD-18-2019
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Patient Satisfaction
Keywords: PCS
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anesthetist controlled group (Other): 15 patients undergoing cataract surgery will receive sedation given by the anesthetist together with local anesthesia according to the depth of sedation in the form of intravenous Midazolam and Fentanyl.
  Interventions: Drug: Midazolam-Fentanyl combination
- Patient-controlled group (Other): 15 patients undergoing cataract surgery under local anesthesia will administer sedation to themselves through a pump.
  Interventions: Drug: Midazolam-Fentanyl combination

INTERVENTIONS:
Drug: Midazolam-Fentanyl combination — Sedation is given to patients undergoing cataract surgery under local anesthesia

SUMMARY:
Perioperative anxiety has many hazards and should be eliminated. Patients undergoing ophthalmologic procedures often undergo it under local anesthesia. In a trial to improve patients' satisfaction sedation is given. Sedation could be given either by an anesthetist or patient-controlled methods. This study compared both methods of sedation in terms of safety, depth of sedation, and patient satisfaction.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted in Kasr Al Ainy Hospital, Ophthalmology surgeries operation theatre, Cairo University, Cairo, Egypt.

After the approval of the research ethical committee (approval number MD-18-2019) & obtaining written informed consent from every patient, 30 patients belonging to the American society of anesthesiologists (ASA) status I, II, aging from 40 to 65 years old, both genders, co-operative patients aware of the instructions, scheduled for cataract surgery under local anesthesia were enrolled for this randomized controlled trial.

However, patients with a diagnosis of cognitive impairment or mental disorder, hypersensitivity to any of the used drugs, having any conditions contraindicating local anesthesia (e.g. Coagulation disorders) were excluded from the study.

Furthermore, patients having severe pulmonary disease e.g. (obstructive sleep apnea), patients using sedative medications within the previous month, and patients with chronic renal and cardiac disorder (e.g. chronic renal failure, heart failure) were also excluded from the study.

Patients were randomly assigned into two equal groups of 15 patients each, the anesthetist controlled group Ga (n=15) and the patient-controlled group Gp (n=15). Randomization was done using computer-generated numbers and the allocation sequence of the participants was concealed in sequentially numbered sealed opaque envelopes.

In the anesthetist controlled group Ga (n=15):

Routine preoperative assessment (proper history taking, examination, and laboratory investigations) was done to all patients as needed.

In the preoperative preparation room, intravenous access (20 gauge cannula) was obtained, premedications were given in the form of (Granitryl at a dose of 10 mcg/kg as an antiemetic and ranitidine at a dose of 0.2 mg/kg as antistress ulcer prophylaxis, they were given diluted with 0.9% sodium chloride solution over 10 minutes), 15 minutes before giving the local anesthesia. Then patients were transferred to the operating room.

In the operating room, all patients were monitored with continuous pulse oximetry, electrocardiogram, and non-invasive blood pressure measured at 10 minutes interval (the blood pressure cuff was applied on the contralateral side of the IV cannula), and oxygen support was given through nasal cannula applied near the nostrils at a flow of 5 liters per minute.

The IV sedation was started before the administration of the local anesthesia in the form of a bolus of 0.02 mg/kg of midazolam and 0.2 mcg/kg of fentanyl to all patients.

Then further doses were given as needed through the procedure according to the depth of sedation. The depth of sedation was assessed at regular intervals (every 10 minutes) using the sedation scale.

A depth of sedation level II or III on the sedation scale was targeted, level I was considered anxious and needs further doses, and more than level III was considered a risk of oversedation.

A soluset was filled with a mixture of 10 mg of midazolam and 150 mcg of fentanyl diluted with 0.9 % sodium chloride solution to complete a total volume of 50 ml. and a concentration of 0.2 mg/ml of midazolam and 3 mcg/ml of fentanyl.

The anesthetist withdrew 2 ml from the soluset and gave them to the patient according to depth of sedation.

In the patient-controlled group Gp (n=15):

Routine preoperative assessment (proper history taking, examination, and laboratory investigations) was done to all patients as needed.

In the preoperative preparation room, intravenous access (20 gauge cannula) was obtained, premedications were given in the form of (Granitryl at a dose of 10 mcg/kg as an antiemetic and ranitidine at a dose of 0.2 mg/kg as antistress ulcer prophylaxis, they were given diluted with 0.9% sodium chloride solution over 10 minutes), 15 minutes before giving the local anesthesia. Then patients were transferred to the operating room.

In the operating room, all patients were monitored with continuous pulse oximetry, electrocardiogram, and non-invasive blood pressure measured at 10 minutes interval (the blood pressure cuff was applied on the contralateral side of the IV cannula), and oxygen support was given through nasal cannula applied near the nostrils at a flow of 5 liters per minute.

The IV sedation was started before the administration of the local anesthesia in the form of a bolus of 0.02 mg/kg of midazolam and 0.2 mcg/kg of fentanyl to all patients.

Patients were instructed on how to use the PCS pump, then the pump (Accufuser) was connected to the IV cannula, patients were given the press button of the infusion pump in one hand and a clicker in the other hand.

Patients were instructed to press the button as often as they feel the need to do so, as there was a lockout interval of six minutes to limit the amount of medication, during this interval the pump will not deliver drugs regardless of the patient's attempts to press the button. The attending anesthetist was instructed to respond to the patient's question "how often should I press the button" with the answer "when you feel unsedated, anxious, irritable, not calm, afraid of the operation and you want to be more relaxed and calm just press the button". If the patient pressed the button during the permission time (after the 6 min lock-out interval), a 2 ml infusion of the drug mixture was administered IV, Otherwise, no drug was administered to the patient.

In this group, patients received a clicker, on the other hand, to press on both the pump and clicker together, every time he/she used the pump to denote the number of attempts.

The observing anesthetist present beside the patient used a stopwatch to record the time from the start of the use of the pump, and the number of the attempts that were recorded as the number of the clicks done by the patient, and so in that way the anesthetist differentiated a true attempt from a false one done during the lockout interval that was fixed at 6 minutes.

The PCS pump was of 100 ml volume, of 2 ml demand doses, 6 minutes lockout interval and of no basal rate of infusion, it was filled with a mixture of 10 mg of midazolam and 150 mcg of fentanyl diluted with 0.9 % sodium chloride solution to complete a total volume of 50 ml. and a concentration of 0.2 mg/ml of midazolam and 3 mcg/ml of fentanyl.

A demand dose of 2 ml with 6 minutes lockout time was used. The patient was unaware of the lockout period, the attending anesthetist was aware of the drug regimen to be present to intervene for adverse events.

Instruction on the use of commercially available PCS pump was given verbally by the anesthetist on the day of surgery and reinforced again in the operation room (OR).

A depth of sedation level II or III on the sedation scale was targeted, level I was considered anxious and needs further doses, and more than level III was considered a risk of oversedation.

In both groups:

The eye to be operated on was marked prior to starting the local anesthesia. The total volume of 8 ml was prepared for the peribulbar block including a mixture of 4 ml lidocaine 2%, 4 ml bupivacaine 0.5%, and 75 IU of hyaluronidase. The anesthetic solution was injected into the extraconal compartment of the eye using two 23 gauge needles with 5 ml being injected at the junction of outer one-third and inner two-thirds of the lower orbital rim and 3 ml were injected superonasally beneath the superior orbital notch. The success of the block was assessed by globe bulge, loss of ocular movements and the eye was padded 5 to 10 minutes (with intermittent pressing 5 seconds and relieve the press for 10 seconds) to enhance the spread of the anesthetic solution and prevent a rise in the intraocular pressure.

After adequate and complete muscle paralysis (assessed by the inability to move the eye in 6 directions known as a gaze), the surgical procedure was allowed by an expert surgeon.

Heart rate, blood pressure, arterial oxygen saturation, and respiratory rate were recorded as a baseline before sedation and at 10 minutes intervals.

Patients' and surgeons' satisfaction, depth of sedation, and patients' anxiety were assessed.

The OR was equipped with emergency equipment and drugs. All the equipment necessary for transformation to general anesthesia if needed at any point were also present including (analgesic, hypnotic, muscle relaxant, laryngoscope, different endotracheal tube sizes a supraglottic device, and a well-functioning anesthesia machine). This transformation would have been needed if a safety endpoint was reached.

Safety endpoints for anesthetist intervention included arterial desaturation < 90%, for more than one minute, hypotension < 90 mmHg systolic or 20% decrease from baseline persisting when repeating determination one minute later, inability to tolerate the procedure, oversedation, airway obstruction, and the need for general anesthesia where the anesthetist will intervene.

At the end of the procedure, the total amount of sedating drug administered was recorded, as well as the number of attempts of self-administration was recorded before discharge from the OR. The patient was transferred to the recovery room and the time to ambulation was calculated, before being discharged to the ward safely.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II.
* Age group 40-65 years old.
* Co-operative patients aware of the instructions.

Exclusion Criteria:

* Diagnosis of cognitive impairment or mental disorder.
* Hypersensitivity to any of the used drugs.
* Contraindication to local anesthesia e.g. Coagulation disorder.
* Severe pulmonary disease e.g. (obstructive sleep apnea).
* Use of sedative medications within the previous month.
* Chronic renal and cardiac disorder e.g. (chronic renal failure, heart failure).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction assessed by 7 point Likert scale. | Intraoperative for 1 hour.
  Assessed by 7 point Likert scale (ranging from 1 as minimum value and 7 as maximal value), higher value is better.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressures. | Intraoperative for 1 hour.
  Measured in mmHg.
Surgeons' satisfaction assessed by 7 point Likert scale. | Intraoperative for 1 hour.
  Assessed by 7 point Likert scale (ranging from 1 as minimum value and 7 as maximal value), higher values are better.
Patient's anxiety assessed by State trait anxiety inventory. | Intraoperative for 1 hour.
  Pre and postoperative, assessed by State-trait anxiety inventory ( a questionnaire of 40 questions), the value is according to patient's answers to the questions.
Heart rate. | Intraoperative for 1 hour.
  Measured in beats per minute.
Oxygen saturation. | Intraoperative for 1 hour.
  In percentage.
Respiratory rate. | Intraoperative for 1 hour.
  In breath per minute.
Time to patient ambulation in minutes. | Postoperative for up to 1 hour.
  The time from end of procedure till the patient is safely discharged from the recovery room, higher values means there is a risk of oversedation which is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Medicine Kasr Al-Ainy Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No